CLINICAL TRIAL: NCT05804188
Title: CRICKET: Critical Events in Anaesthetised Kids Undergoing Tracheal Intubation
Acronym: CRICKET
Status: Recruiting | Type: Observational
Sponsor: Thomas Riva (Other)
Collaborators: University of Bern (Other); The Hospital for Sick Children (Other); Boston Childrenâ€™s Hospital (Unknown); Istituto Giannina Gaslini (Other)
Responsible Party: Sponsor-Investigator, Thomas Riva, Prof. Dr. med., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: Cricket 2023; 2023-00246 (Registry Identifier: Swissethics)
Record Dates: First submitted 2023-03-23; First posted 2023-04-07 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Intubation Complication; Adverse Events
Keywords: Intubation, Intratracheal; Anesthesiology; Difficult Airway; Critical events; Pediatrics
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: tracheal intubation — children between 0-16 requiring tracheal intubation

SUMMARY:
The investigators' overall objective is to assess the incidence of critical events related to tracheal intubation at all international study sites. Furthermore, the study will investigate the used intubation techniques and identify possible improvement measures to increase patient safety.

DETAILED DESCRIPTION:
It is a prospective observational multi-centre study collecting health related patient data over a period of three months. This serves best the study's purpose to detect the incidence and nature of problems related to tracheal intubation and how such problems are handled with the aim to further improve patient safety. During the observational period the anaesthesia staff in charge will complete a screening questionnaire for critical events associated with tracheal intubation for every patient undergoing general anaesthesia with tracheal intubation. If no critical events arise there are no further requirements. If a critical event occurs, the anaesthesia provider will complete a more detailed questionnaire which includes more questions about what exactly happened.

Patient characteristics will be extracted from the anaesthesia records. The investigators will extract such data for all patients undergoing tracheal intubation and additional data for those with critical events. The research will not intervene with the clinical conduct of patient care.

The collected health related data will be transferred to an electronic research data base. In this data base data will be encoded. Every patient with a critical event will be followed up as described above.

ELIGIBILITY:
Inclusion Criteria:

* All paediatric patients requiring tracheal intubation, performed by the anaesthesia team for procedures or interventions requiring general anaesthesia
* Patients from 0 - 16 years of age.
* Informed or general consent given, according to the relevant ethics committee statement.

Exclusion Criteria:

* Refusal to give consent or withdrawal of consent if such is required by the relevant ethics committee.
* Patients >16 years

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All paediatric patients requiring tracheal intubation due to their medical condition are screened if they fulfill the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 105000 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with critical events related to intubation | Maximum of 30 days
  Primary study outcome is the incidence of anaesthesia cases with critical events associated with endotracheal intubation requiring intervention from the start of anaesthesia until the discharge of the patient from the post-anaesthesia care unit or end of anaesthesia (defined as handover to the paediatric or neonatal intensive care unit, the ward or discharge home straight from anaesthesia care) in children aged 0 - 16 years. Facultatively for those who do not have capacity the acquisition of data stops at the end of anaesthesia (defined as handover to the post-anaesthesia care unit).

SECONDARY OUTCOMES:
Number of patients with severe hypoxemia | 1 hour
  Oxygen saturation (SpO2) < 85% or >20 points below initial value at least 60 seconds
Number of patients with severe bradycardia | 1 hour
  0-3 months old: Heart rate (HR) < 80 bpm
  * 4 months - 2 years: HR < 60 bpm
  * 2-10 years old: HR < 40 bpm
  * 10-16 years old: HR < 30 bpm at least 1 minute
Number of patients with esophageal intubation | 1 hour
  Tracheal tube placed in the oesophagus diagnosed by (video-) laryngoscopy, absence of sustained end-tidal carbon dioxide (EtCO2) trace, absence of lung ventilation (auscultation or absence of chest excursions) causing a drop in oxygenation
Number of patients with laryngospasm | 1 hour
  Complete airway obstruction associated with rigidity of the abdominal and chest walls and leading to unsuccessful child's ventilation, or glottic closure associated with chest movement but silent unsuccessful child's respiratory efforts and assisted ventilation, unrelieved in both situations with simple jaw thrust and continuous positive airway pressure (CPAP) manoeuvres and requiring the administration of medication (propofol, suxamethonium etc.) and/or tracheal (re)-intubation
Number of patients with bronchospasm | 1 hour
  Increased respiratory effort, especially during expiration, and wheeze on auscultation. Episode of bronchospasm requires the administration of a bronchodilator.
Number of patients with stridor after extubation | 1 hour
  Severe inspiratory flow limitation with sternal retraction, intrathoracic pressure swing, and potentially cyanosis occurring after extubation with or without the administration of oxygen, intravenous steroids and/or epinephrine (nebulization) or tracheal intubation. This can be documented clinically or with diagnostic examination, with persistence of symptoms.
Number of patients with obstruction of tracheal tube | 1 hour
  Obstruction of tracheal tube needing lavage or tube exchange
Number of patients with airway bleeding | 1 hour
  Acute bleeding from nose, arytenoids or pharynx causing obstruction or risk for pulmonary aspiration
Number of patients with can't intubate, can't oxygenate (CICO) situation | 1 hour
  Situation when there is failed intubation and failure to adequately oxygenate using facemask ventilation or supraglottic airway device resulting in increasing hypoxemia in an anaesthetised and paralysed patient
Number of patients with severe bradycardia/Cardiac arrest | 1 hour
  Cessation of circulation (no pulse) or severe bradycardia (i.e. fibrillation/tachycardia) requiring chest compressions, during the intubation/extubation manoeuvres.
Number of patients with pulmonary aspiration | 1 hour
  Presence of non-respiratory secretions (gastric, particulate, blood) in the airway as evidenced by (video-) laryngoscopy, suctioning, or bronchoscopy or radiologic signs.
Number of patients with pneumothorax/ pneumomediastinum | 1 hour
  Air in the thorax and/or mediastinum as consequence of tracheal intubation and ventilation, causing lung collapse or mediastinum dislodgment diagnosed by Lung-ultrasound and/or X-ray.
Number of patients with negative pulmonary oedema | 1 hour
  Non-cardiogenic pulmonary oedema that results from the generation of high negative intrathoracic pressure needed to overcome upper airway obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD, Prof, Study Chair — Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University
Locations (8):
- United States (2):
  - Department of Anesthesiology, Critical Care and Pain Medicine, Boston, Massachusetts
  - Dept of Anesthesiology and Critical Care Medicine, The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Department of Anaesthesia and Pain Management, Perth Children's Hospital, Perth, Australia
- Canada (2):
  - Dept. Anesthesia, The Hospital for Sick Children, Toronto, Ontario
  - Dept. Anesthesia, Montreal Children's Hospital, McGill University Health Centre, Montreal
- Department of Cardiac Anesthesiology and Intensive Care Medicine, Charité Universitätsmedizin, Berlin, Germany
- Switzerland (2):
  - Children's Hospital Zurich, Zurich, Canton of Zurich
  - Unité d'anesthésie pédiatrique, Hôpital des Enfants / HUG, Geneva

IPD SHARING:
Plan to Share IPD: No